CLINICAL TRIAL: NCT01672242
Title: Assessment of End Expiratory Lung Volumes in Healthy Subjects Using High Flow Oxygen (Vapotherm®)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Maryland, Baltimore (Other)
Collaborators: Vapotherm, Inc. (Industry)
Responsible Party: Principal Investigator, Carl Shanholtz, Professor of Medicine, University of Maryland, Baltimore
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: HP-00052656
Record Dates: First submitted 2012-08-09; First posted 2012-08-24 (Estimated); Results first posted 2018-01-10 (Actual); Last update posted 2022-03-08 (Actual); Status verified 2022-03

CONDITIONS: Healthy Adult Volunteers
MeSH Terms: interventions — Continuous Positive Airway Pressure

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- HFNC (Experimental): High Flow Nasal Cannula (HFNC) oxygen.
  Interventions: Device: HFNC
- CPAP (Experimental): Continuous Positive Airway Pressure (CPAP)
  Interventions: Device: CPAP

INTERVENTIONS:
Device: HFNC — Graded high flow nasal cannula oxygen at 10, 20 , 30, and 40 liters per minute (LPM) to each subject and end-expiratory lung volume measured by respiratory inductive plethysmography.
  Other Names: High flow nasal cannula oxygen, Precision Flow®, Vapotherm®
  Arms: HFNC
Device: CPAP — Graded contiuous positive airway pressure at 5, 10 , 15, and 20 cm H2O applied to each subject and end-expiratory lung volume measured by respiratory inductive plethysmography.
  Other Names: Continuous positive airway pressure, Respironics(R)
  Arms: CPAP

SUMMARY:
Respiratory distress is a common problem in an intensive care unit. There are multiple mechanisms that are used to help patients who are in respiratory distress including mechanical ventilation, continuous positive airway pressure (CPAP), bilevel positive airway pressure (BiPAP), high flow oxygen, and oxygen supplementation through nasal cannula or a facemask.

The purpose of this study is to evaluate the mechanism by which Vapotherm, a high flow oxygen system, provides breathing support. Vapotherm provides high flow oxygen at different flow rates, meaning one can increase the amount of oxygen flow to help with breathing support. The investigators believe that this high flow oxygen system may provide similar breathing support that a continuous positive airway pressure machine (CPAP) machine does.

DETAILED DESCRIPTION:
High flow nasal cannula oxygen therapy (HFNC) is a method of oxygen delivery now commonly used in persistently hypoxic patients refractory to conventional modes of oxygen supplementation (i.e. nasal cannula, facemask, non-rebreather facemask). Initially used in neonates, it is now increasingly popular in the adult population. While the investigators know how HFNC provides oxygen supplementation, the physiologic mechanism of correcting hypoxemia is still unclear. There are five mechanisms of hypoxemia, four which correct with oxygen supplementation - decreased fraction of inspired oxygen (FiO2), hyperventilation, ventilation-perfusion (V/Q) mismatch, and diffusion defect; and one that does not - shunt. The hypoxemia refractory to supplemental oxygen suggests the presence of physiologic shunt. The conventional non-invasive therapy to reduce shunt fraction requires raising end-expiratory lung volumes by raising end-expiratory airway pressures using the application of continuous positive airway pressure (CPAP) or bilevel positive airway pressure (BiPAP). The Vapotherm® (Vapotherm®, Stevensville, Maryland) product of high flow oxygen therapy (Precision Flow®) is one the investigators frequently use in intensive care units at the University of Maryland Medical Center. It does not create a leak proof seal in the nose as seen in CPAP and BiPAP. Positive pressure generation has been studied in another high flow oxygen system called Optiflow™ (Fisher & Paykel Healthcare, Ltd., Auckland, New Zealand). However this device differs from Vapotherm® in that its nasal bores are large and create a seal in each nares thereby affected both ventilation and the level of positive end expiratory pressure (PEEP) generation. Additionally, these studies measured positive expiratory lung pressures, not volume. Positive end expiratory alveolar pressure and increase expiratory lung volumes in adults have not yet been demonstrated using Precision Flow®.

HFNC is intriguing because studies and clinical data have shown it is a relatively non-invasive method of oxygen delivery that appears to correct hypoxemia better than other non-invasive methods. It is more comfortable than a CPAP machine and thus is better tolerated among patients, especially those who are critically ill and possibly altered. While it has been used in neonates for some time, its use with adults is new and needs more research.

The investigators hypothesis is that HFNC corrects persistent hypoxemia by producing increased end-expiratory lung volumes thus keeping alveoli open throughout the respiratory cycle which other oxygen supplements are unable to do. Using healthy volunteers the investigators will measure end expiratory lung volumes on HFNC and compare them to those obtained with CPAP at graded pressures.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 75
* Able to follow and understand simple instructions to collect spirometry

Exclusion Criteria:

* Younger than 18y/o
* Older than 75 years old
* History of chronic obstructive pulmonary disease (COPD)
* History of asthma
* History of congestive heart failure
* Measured ratio of forced expiratory volume at 1 second/forced vital capacity (FEV1/FVC) <70 when undergoing spirometry

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2012-07; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Carl B. Shanholtz, MD, Principal Investigator — University of Maryland
Locations (1):
- University of Maryland School of Medicine, Baltimore, Maryland, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Normal subjects were recruited from the University of Maryland School of Medicine
Pre-assignment Details: Volunteers were asked briefly about their health status and given spirometry to document no evidence of obstructive airways disease or other chronic lung disease that would impact their FRC measurements with high flow nasal cannula therapy or CPAP.
Groups:
- HFNC-CPAP: High flow nasal cannula oxygen first period, followed by continuous positive airway pressure second period.
- CPAP-HFNC: Continuous Positive Airway Pressure first period, followed by high flow nasal cannula second period.
Period: Period 1
Arm/Group | HFNC-CPAP | CPAP-HFNC
Started | 4 | 2
Completed | 4 | 2
Not Completed | 0 | 0
Period: Period 2
Arm/Group | HFNC-CPAP | CPAP-HFNC
Started | 4 | 2
Completed | 4 | 2
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Normal healthy adult volunteers
Groups:
- Participants: Normal healthy adult volunteers
Arm/Group | Participants
Number analyzed (Participants) | 6
Age, Continuous [Median (Inter-Quartile Range); unit: years] — Age
  years | 35.5 [32.75 to 56]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 6
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 6
height [Median (Inter-Quartile Range); unit: inches] | 71 [68.5 to 74]
predicted body weight [Median (Inter-Quartile Range); unit: kg] | 75.3 [68.4 to 82.2]
FEV1 (% predicted) [Median (Inter-Quartile Range); unit: % predicted] | 93 [90 to 102]
FEV1/FVC (%) [Median (Inter-Quartile Range); unit: ratio] | 102 [97 to 107]

OUTCOME MEASURES:

1. Primary Outcome: Change in End-expiratory Lung Volume
Description: Change in end-expiratory lung volume from baseline arbitrarily set at 0 mL.
Time Frame: baseline and after 3-5 minutes after each level of flow or pressure
Measure: Mean (Standard Deviation); unit: mL
Groups:
- HFNC: High flow nasal cannula oxygen 40 liters/min
- CPAP: Continuous positive airway pressure 20 cm H2O
Arm/Group | HFNC | CPAP
Number analyzed (Participants) | 6 | 6
mL | -144 (317) | 103 (274)

ADVERSE EVENTS:
Time Frame: 6 hours
Groups:
- HFNC: High flow nasal cannula
- CPAP: Continuous positive airway pressure
Arm/Group | HFNC | CPAP
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/6
Other Adverse Events (participants affected / at risk) | 0/6 | 0/6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No